CLINICAL TRIAL: NCT01940172
Title: A Phase 1b, Open-label, Non-randomized Multicenter Study of Birinapant in Combination With Conatumumab in Subjects With Relapsed Epithelial Ovarian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer
Brief Title: Study of Birinapant in Combination With Conatumumab in Subjects With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL32711-POC-0090-PTL
Record Dates: First submitted 2013-09-06; First posted 2013-09-12 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Relapsed Epithelial Ovarian Cancer; Relapsed Primary Peritoneal Cancer; Relapsed Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — birinapant; conatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Birinapant with Conatumumab (Experimental)
  Interventions: Drug: Birinapant; Drug: Conatumumab

INTERVENTIONS:
Drug: Birinapant — Dose Escalation:
  Dose Level (1) - 13 mg/m2 (twice a week for 3 of 4 weeks); Dose Level (-1) - 11 mg/m2 (twice a week for 3 of 4 weeks); Dose Level (2) - 13 mg/m2 (twice weekly for 4 weeks );
  Other Names: TL32711
Drug: Conatumumab — 10 mg/kg IV on Day 1 and 15 of each cycle

SUMMARY:
This is a dose escalation study in female subjects with relapsed ovarian cancer (including epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer). Approximately 30 to 40 subjects will be administered a combination of conatumumab and birinapant.

In the initial dose-escalation stage of the study, adult female subjects will receive conatumumab in combination with increasing doses of birinapant in dose-escalation cohorts to determine the MTD of birinapant when administered with a fixed dose of conatumumab.

In safety expansion stage, adult female subjects will receive conatumumab in combination with birinapant at the MTD of the combination.

ELIGIBILITY:
Inclusion Criteria-If subject:

* Is a women who is at least 18 years of age.
* Has a negative serum pregnancy test at screening for women of childbearing potential.
* Pathologically confirmed ovarian cancer (epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer) may have had a maximum of 3 prior systemic chemotherapy regimens (excluding hormonal therapies and investigational agents).
* Has a performance status of 0 or 1 by the Eastern Cooperative Oncology Group (ECOG) scale.
* Has a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria AND meet Gynecologic Cancer InterGroup (GCIG) CA 125 criteria.
* Has a life expectancy of at least 3 months.
* Has adequate liver, renal, pancreatic, coagulation and bone marrow function.

Exclusion Criteria-If subject:

* Has symptomatic or uncontrolled brain metastases requiring current treatment (<8 weeks from last cranial radiation treatment or <4 weeks from last steroid treatment).
* Has known intolerance to any of the study drugs or any of their excipients.
* Has known or suspected diagnosis of human immunodeficiency virus (HIV) or chronic active Hepatitis B or C.
* Has uncontrolled hypertension defined as blood pressure >160/100 mmHg without medication, or not controlled despite medications.
* Has received systemic chemotherapy, hormonal therapy, immunotherapy, anti-tumor necrosis factor (TNF) therapies, experimental or approved anticancer proteins/antibodies therapy

  ≤28 days before enrollment.
* Has impaired cardiac function or clinically significant cardiac disease including the following:

  1. New York Heart Association Grade III or IV congestive heart failure.
  2. Myocardial infarction within the last 12 months prior to dosing with birinapant.
* Has a QT interval corrected for heart rate (QTcB) >480 msec (including subjects on medication). Subjects with a ventricular pacemaker for whom QT interval is not measurable may be eligible.
* Has a lack of recovery of prior adverse non-hematological events to Grade ≤1 severity (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.03) (except alopecia) due to therapy administered prior to the initiation of study drug dosing.
* Has any concurrent disease and/or medical condition that, in the opinion of the Investigator, would prevent the subject's participation, render the subject at excessive risk (including excessive risks due to the toxicity profile of the planned combination chemotherapeutic regimen), or limit the subject's compliance with the protocol's required evaluations.
* Has a prior history of cranial nerve palsy.
* Has autoimmune diseases or inflammatory diseases, for example, active rheumatoid arthritis, active inflammatory bowel disease or any chronic inflammatory conditions.
* Has pseudomyxoma, mesothelioma, unknown primary tumor, sarcoma, neuroendocrine histology, clear cell or mucinous histology or subjects with borderline ovarian cancer.
* Requires concomitant chronic use of anti-TNF therapies, corticosteroids or nonsteroidal anti- inflammatory drugs (NSAIDS). Intermittent use (7 or fewer days per 14 days) of corticosteroids as pre-medications is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) | 28 Days

SECONDARY OUTCOMES:
Clinical response as measured by RECIST (v1.1) criteria, CA 125 (GCIG criteria) and progression-free survival (PFS). | Up to 4 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - TetraLogic research site, Fresno, California
  - TetraLogic Research Site, San Luis Obispo, California
  - TetraLogic Research Site, Fairway, Kansas
  - TetraLogic Research Site, Boston, Massachusetts
  - TetraLogic Research Site, Durham, North Carolina
  - TetraLogic Research Site, Philadelphia, Pennsylvania
  - TetraLogic Research Site, Nashville, Tennessee
  - TetraLogic Research Facility, Dallas, Texas